CLINICAL TRIAL: NCT06971393
Title: A Comparison of Health Literacy Estimates Among Patients, Caregivers and a Geriatric Team
Brief Title: Health Literacy in Geriatric Patients
Status: Recruiting | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Christopher Patterson, Principal Investigator, Hamilton Health Sciences Corporation
Other Study IDs: 17823
Record Dates: First submitted 2024-12-08; First posted 2025-05-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-12

CONDITIONS: Health Literacy
Keywords: Health Literacy; Geriatric health literacy assessment; Health literacy in tertiary care settings; Correlation of health literacy and health outcomes; BRIEF health literacy questionnaire; Visual Analogue Scale quality of life measure; Emergency room visits and hospitalization tracking in geriatric population; Patient-provider health literacy perception agreement; Patient, caregiver, and geriatric team health literacy alignment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Health Literacy is one's ability to understand health information well enough to make informed decisions about their health. Limited health literacy makes it hard for people to understand complex health issues and follow health care recommendations. Limited health literacy is associated with adverse health outcomes such as higher mortality, increased risk of emergency department visits and hospital admissions leading to higher medical costs. Although there are tools to assess health literacy, they are not widely used, so many healthcare providers do not measure their patients' health literacy levels adequately. Health care workers tend to overestimate their patients' health literacy. This is especially important for older adults who often have memory problems and multiple illnesses. This study will evaluate how doctors and team members in a geriatric clinic estimate their patient's health literacy and determine if this matches with the patients' health literacy as measured by a simple validated questionnaire. The investigators will also look at how a patient's relative or caregiver estimates their health literacy using a similar short questionnaire. The research team plans to follow up with a telephone call in 6 months, to see which health concerns if any have occurred since the clinic visit.

DETAILED DESCRIPTION:
As treatments become more sophisticated and the healthcare system becomes more complex, health literacy (HL) assumes an ever-greater importance in the therapeutic alliance between healthcare professionals and patients.

Limited health literacy causes difficulty in understanding one's health condition. As a result, it is associated with less adherence to self-care behaviours, increased mortality, increased hospitalizations, other adverse health outcomes, and high healthcare costs. In those over aged 65, health literacy is positively influenced by levels of educational attainment and literacy practices in the home, male gender, and weakly by informal learning and self-study and adult education experience. Negative associations include being foreign-born and failure to learn from exposure to various contexts. Understanding the health literacy of patients is particularly vital for geriatricians as older adults referred to geriatric medicine clinics already experience barriers to high quality care due to the frequent presence of cognitive impairment and multiple comorbidities.

The interaction among these variables and health literacy in a tertiary care setting for older adults with cognitive impairment remains under-explored. Given the dependent state of many cognitively impaired individuals, the responsibility lies with geriatricians to adjust their communication and care strategies according to the HL levels of their patients. Studying the association between the accuracy of geriatrician-perceived HL and health outcomes could reveal the extent to which physician communication impacts these outcomes. Given these intertwined factors, a 6-month follow-up is crucial to capture the longitudinal associations of HL on patient outcomes, providing a more comprehensive picture of how these variables interact over time.

This study's primary outcome is the evaluation of patient health literacy and the level of agreement between the geriatric team's perception and objectively measured health literacy. The secondary outcome is assessing how patient health literacy is associated with medication adherence and future planning. As well, the investigators hope to assess how patient health literacy is associated with emergency department visits, hospitalizations, hospital length of stay, remaining home, long-term care admission and mortality within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients (both new and follow up) attending St. Peter's Hospital Geriatric Clinic
* Willingness to participate in the study (caregiver can rate HL for patient if patient unable to)
* Consenting to study (by patient or caregiver)

Exclusion Criteria:

* Behavior (e.g. behavioral and psychological symptoms of dementia) which may be aggravated by additional questions
* Acute illness preventing participation
* Terminal illness that would prevent 6-month telephone follow up
* Previous participation in this study

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who have been referred by their primary care or other physicians, to the Geriatric Clinic at the St. Peter's Hospital site of Hamilton Health Sciences Corporation. All patients, including new referrals and follow up patients will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient self-identified HL | At enrollment
  The patient's self-identified health literacy based on the BRIEF, a 4-item measure of health literacy that has been validated for older adults.
Caregiver's perception of patient's HL | At enrollment
  The caregiver's perception of the patient's health literacy based on the BRIEF-C, a tool based on the BRIEF, constructed to reflect the caregiver's perception of the patient's HL.
Patient self-identified quality of life | At enrollment
  The patient's self-identified quality of life measured by the EQ-VAS, a visual analogue scale measuring quality of life on a scale of 0 to 100
Geriatric Team's assessment of patient's HL | At enrollment
  Geriatric Team will report HL as Adequate/marginal/inadequate. Level of adequacy (1,2,3) is optional

SECONDARY OUTCOMES:
Medication adherence | At enrollment
  Low medication adherence is predictive of poor health outcomes for older adults and is associated with education level, health literacy, patient satisfaction, and sufficient communication. However, associations have not been delineated in an outpatient setting or using a validated HL scale.
  Adherence will be measured by dichotomous outcome (80% adherent vs non-adherent) according to the consultation note.
Number of participants with existing community home care planning | At enrollment
  Home and community care includes access to long-term or short-term nursing, home support, and other services. As well, the use of these services has a significant effect on healthy aging in place. However, it is currently unknown the extent to which HL may influence an individual's ability to obtain home care.
Number of participants with long-term care planning | At enrollment
  Long term care planning includes discussion about or application to long term care facility admission.
Number of patients with code status discussion | At enrollment
  Statement about advance directives or POST in medical record.
Power of Attorney designation | At enrollment
  Whether a patient has discussed and identified a power of attorney.
Number of patients remaining home | At enrollment
  Whether the patient is living in community residence
Falls | At enrollment
  Number of Falls in the past year
Number of ED visits | 6 months
  Number of ED visits during follow up period (6 months)
Number of hospitalizations | 6 months
  Number of hospital admissions during follow up period (6 months)
Hospital length of stay | 6 months
  Number of days patient admitted to hospital during follow up period (6 months)
Long-term care admission | 6 months
  Whether the patient was admitted to long-term care at follow up
Mortality | 6 months
  Whether patient died during the follow up period (6 months)
Injurious Falls | 6 months
  Frequency of falls experienced by the patient before the follow up period.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Peter's Geriatric Clinic, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD for this health literacy study will not be shared in order to protect participant privacy and maintain confidentiality, given the sensitivity of the data related to personal health literacy levels, caregiver insights, and healthcare team perceptions.

REFERENCES:
- [Background] Kobayashi LC, Wardle J, von Wagner C. Internet use, social engagement and health literacy decline during ageing in a longitudinal cohort of older English adults. J Epidemiol Community Health. 2015 Mar;69(3):278-83. doi: 10.1136/jech-2014-204733. Epub 2014 Nov 26. PMID 25428933
- [Background] Chesser AK, Keene Woods N, Smothers K, Rogers N. Health Literacy and Older Adults: A Systematic Review. Gerontol Geriatr Med. 2016 Mar 15;2:2333721416630492. doi: 10.1177/2333721416630492. eCollection 2016 Jan-Dec. PMID 28138488
- [Background] Lu J, Sun S, Gu Y, Li H, Fang L, Zhu X, Xu H. Health literacy and health outcomes among older patients suffering from chronic diseases: A moderated mediation model. Front Public Health. 2023 Jan 10;10:1069174. doi: 10.3389/fpubh.2022.1069174. eCollection 2022. PMID 36703841
- [Background] Li H, Tao S, Sun S, Xiao Y, Liu Y. The relationship between health literacy and health-related quality of life in Chinese older adults: a cross-sectional study. Front Public Health. 2024 Mar 20;12:1288906. doi: 10.3389/fpubh.2024.1288906. eCollection 2024. PMID 38572002
- [Background] Geboers B, Uiters E, Reijneveld SA, Jansen CJM, Almansa J, Nooyens ACJ, Verschuren WMM, de Winter AF, Picavet HSJ. Health literacy among older adults is associated with their 10-years' cognitive functioning and decline - the Doetinchem Cohort Study. BMC Geriatr. 2018 Mar 20;18(1):77. doi: 10.1186/s12877-018-0766-7. PMID 29558890
- [Background] Suppiah SD, Malhotra R, Tan YW, Jessup RL, Chew LST, Tang WE, Beauchamp A. Prevalence of health literacy and its correlates from a national survey of older adults. Res Social Adm Pharm. 2023 Jun;19(6):906-912. doi: 10.1016/j.sapharm.2023.02.013. Epub 2023 Feb 27. PMID 36898905
- [Background] Wang Q, Fan K, Li P. Effect of the Use of Home and Community Care Services on the Multidimensional Health of Older Adults. Int J Environ Res Public Health. 2022 Nov 21;19(22):15402. doi: 10.3390/ijerph192215402. PMID 36430119
- [Background] Jin H, Kim Y, Rhie SJ. Factors affecting medication adherence in elderly people. Patient Prefer Adherence. 2016 Oct 19;10:2117-2125. doi: 10.2147/PPA.S118121. eCollection 2016. PMID 27799748
- [Background] Lapid MI, Rummans TA, Boeve BF, McCormick JK, Pankratz VS, Cha RH, Smith GE, Ivnik RJ, Tangalos EG, Petersen RC. What is the quality of life in the oldest old? Int Psychogeriatr. 2011 Aug;23(6):1003-10. doi: 10.1017/S1041610210002462. Epub 2011 Feb 1. PMID 21281556
- [Background] Feng Y, Parkin D, Devlin NJ. Assessing the performance of the EQ-VAS in the NHS PROMs programme. Qual Life Res. 2014 Apr;23(3):977-89. doi: 10.1007/s11136-013-0537-z. Epub 2013 Oct 1. PMID 24081873
- [Background] Shmueli A. The relationship between the visual analog scale and the SF-36 scales in the general population: an update. Med Decis Making. 2004 Jan-Feb;24(1):61-3. doi: 10.1177/0272989X03261562. PMID 15005955
- [Background] Rawson KA, Gunstad J, Hughes J, Spitznagel MB, Potter V, Waechter D, Rosneck J. The METER: a brief, self-administered measure of health literacy. J Gen Intern Med. 2010 Jan;25(1):67-71. doi: 10.1007/s11606-009-1158-7. Epub 2009 Nov 3. PMID 19885705
- [Background] Federman AD, Sano M, Wolf MS, Siu AL, Halm EA. Health literacy and cognitive performance in older adults. J Am Geriatr Soc. 2009 Aug;57(8):1475-80. doi: 10.1111/j.1532-5415.2009.02347.x. Epub 2009 Jun 8. PMID 19515101
- [Background] Sudore RL, Mehta KM, Simonsick EM, Harris TB, Newman AB, Satterfield S, Rosano C, Rooks RN, Rubin SM, Ayonayon HN, Yaffe K. Limited literacy in older people and disparities in health and healthcare access. J Am Geriatr Soc. 2006 May;54(5):770-6. doi: 10.1111/j.1532-5415.2006.00691.x. PMID 16696742
- [Background] Voigt-Barbarowicz M, Brutt AL. The Agreement between Patients' and Healthcare Professionals' Assessment of Patients' Health Literacy-A Systematic Review. Int J Environ Res Public Health. 2020 Mar 31;17(7):2372. doi: 10.3390/ijerph17072372. PMID 32244459
- [Background] Bass PF 3rd, Wilson JF, Griffith CH, Barnett DR. Residents' ability to identify patients with poor literacy skills. Acad Med. 2002 Oct;77(10):1039-41. doi: 10.1097/00001888-200210000-00021. PMID 12377684
- [Background] Tarpila S. [Dietary fiber and health]. Duodecim. 1982;98(22):1738-47. No abstract available. Finnish. PMID 6307631
- [Background] Kelly PA, Haidet P. Physician overestimation of patient literacy: a potential source of health care disparities. Patient Educ Couns. 2007 Apr;66(1):119-22. doi: 10.1016/j.pec.2006.10.007. Epub 2006 Nov 30. PMID 17140758
- [Background] Kim S, Won CW, Kim BS, Kim S, Yoo J, Byun S, Jang HC, Cho BL, Son SJ, Lee JH, Park YS, Choi KM, Kim HJ, Lee SG. EuroQol Visual Analogue Scale (EQ-VAS) as a Predicting Tool for Frailty in Older Korean Adults: The Korean Frailty an Aging Cohort Study (KFACS). J Nutr Health Aging. 2018;22(10):1275-1280. doi: 10.1007/s12603-018-1077-6. PMID 30498837
- [Background] Al Ghassani A, Rababa M. Factors Associated with Home Care Outcomes among Community-Dwelling Older Adult Patients with Dementia. Dement Geriatr Cogn Dis Extra. 2021 May 6;11(2):99-109. doi: 10.1159/000516086. eCollection 2021 May-Aug. PMID 34178013
- [Background] Tan V, Chen C, Merchant RA. Association of social determinants of health with frailty, cognitive impairment, and self-rated health among older adults. PLoS One. 2022 Nov 11;17(11):e0277290. doi: 10.1371/journal.pone.0277290. eCollection 2022. PMID 36367863
- [Background] Eichler K, Wieser S, Brugger U. The costs of limited health literacy: a systematic review. Int J Public Health. 2009;54(5):313-24. doi: 10.1007/s00038-009-0058-2. Epub 2009 Jul 31. PMID 19644651
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Kobayashi LC, Wardle J, Wolf MS, von Wagner C. Aging and Functional Health Literacy: A Systematic Review and Meta-Analysis. J Gerontol B Psychol Sci Soc Sci. 2016 May;71(3):445-57. doi: 10.1093/geronb/gbu161. Epub 2014 Dec 11. PMID 25504637
- [Background] Haun J, Luther S, Dodd V, Donaldson P. Measurement variation across health literacy assessments: implications for assessment selection in research and practice. J Health Commun. 2012;17 Suppl 3:141-59. doi: 10.1080/10810730.2012.712615. PMID 23030567